CLINICAL TRIAL: NCT06874517
Title: Greek vs. Egyptian Foot: The Impact of Second Toe Length on Hallux Valgus Development
Brief Title: Second Toe Length and Hallux Valgus: Greek vs. Egyptian Foot
Status: Recruiting | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: BeylikduzuStateH15
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
A total of 150 patients aged 60-80 years with existing foot radiographs will be included in the study. Radiographic evaluations will include measurements of the hallux valgus angle, first intermetatarsal angle, and the metatarsal and phalanx lengths of the first and second toes. The ratio of the second toe phalanx length to the first toe phalanx length will be calculated and recorded. The relationship between the hallux valgus angle, toe lengths, and their ratios will be analyzed using statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Age between 60-80 years
* Presence of foot radiographs suitable for measurement
* No history of prior foot surgery

Exclusion Criteria:

* History of foot trauma or fractures
* Previous foot or toe surgery
* Presence of congenital foot deformities
* Neurological or rheumatologic conditions affecting foot structure
* Severe osteoarthritis or other degenerative foot diseases visible on radiographs

Ages: 60 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 150 patients aged 60-80 years who have existing foot radiographs suitable for measurement.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Hallux Valgus Angle | 0 day
  The angle between the first metatarsal and the proximal phalanx of the first toe, measured on radiographs. Higher values indicate greater hallux valgus severity.

SECONDARY OUTCOMES:
First Intermetatarsal Angle | 0 day
  The angle between the first and second metatarsal bones, measured on radiographs. Higher values are associated with increased deformity.
First Toe (Hallux) Metatarsal and Phalanx Lengths | 0 day
  The length of the first metatarsal and its phalanges, measured on radiographs.
Second Toe Metatarsal and Phalanx Lengths | 0 day
  The length of the second metatarsal and its phalanges, measured on radiographs.
Second Toe to First Toe Phalanx Length Ratio | 0 day
  The ratio of the second toe phalanx length to the first toe phalanx length, calculated to assess relative toe length differences.

CONTACTS AND LOCATIONS:
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Beylikdüzü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No